CLINICAL TRIAL: NCT00942487
Title: Effects of NEbivolol on Subclinical Left Ventricular dYSfunction. A Comparative Study Against Metoprolol. The ENESYS Study. A Phase 3, Randomised, Parallel, Active-controlled, Open Label Study
Brief Title: Effects of Nebivolol on Subclinical Left Ventricular dySfunction: A Comparative Study Against Metoprolol
Acronym: ENESYS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Berlin-Chemie Menarini (Industry)
Responsible Party: Professor Dragos VINEREANU, University and Emergency Hospital of Bucharest
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MeRo/04/Neb-LVD/003
Record Dates: First submitted 2009-07-19; First posted 2009-07-21 (Estimated); Last update posted 2009-07-21 (Estimated); Status verified 2009-07

CONDITIONS: Primary Arterial Hypertension
Keywords: arterial hypertension
MeSH Terms: conditions — Hypertension | interventions — Nebivolol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nebivolol (Experimental)
  Interventions: Drug: Nebilet
- Metoprolol (Active Comparator)
  Interventions: Drug: Corvitol

INTERVENTIONS:
Drug: Nebilet — Trade-mark: Nebilet® (Berlin-Chemie Menarini) INN: nebivolol Dosage and route of administration: 5 mg tablets, o.d. for oral administration
  Arms: Nebivolol
Drug: Corvitol — Trade-mark: Corvitol (Berlin-Chemie Menarini) INN: metoprolol Dosage and route of administration: 50 mg tablets, b.d. (100 mg/day) for oral administration
  Arms: Metoprolol

SUMMARY:
Summary:

* Study title: Effects of Nebivolol on subclinical left ventricular dysfunction. A comparative study against Metoprolol. (ENESYS study)
* Study phase: 3
* Study design (parallel, cross-over, etc.), randomisation and blinding procedures, type of control (placebo or active): randomised, parallel, active-controlled, open label
* Study treatment(s)/drug(s): Nebivolol versus Metoprolol
* Patients:

  * characteristics: patients with hypertension and left ventricular hypertrophy
  * planned total number: 50
* Study duration:

  * total enrolment period (months): 18
  * treatment period (months): 6
  * follow up period (months): 6
* Total study duration (months): 24

  * Number of Centres: 1
  * Country(ies): Romania (RO)

DETAILED DESCRIPTION:
STUDY OBJECTIVES

1. PRIMARY:

   * Longitudinal myocardial velocities at rest (assessed by tissue Doppler echocardiography)
   * Systolic functional reserve (calculated as the absolute and relative increase of the myocardial systolic velocities at peak stress from rest)
   * Brain natriuretic peptide (BNP, NT-pro BNP) after a 6-months period of treatment with nebivolol versus metoprolol. An improvement of more than 20% of the myocardial resting velocities of systolic functional reserve is considered to be clinically relevant. The working hypothesis is that the improvement of subclinical left ventricular dysfunction after 6 months of treatment is going to be greater in patients who receive nebivolol than in those who receive metoprolol.
2. SECONDARY:

   * Global systolic function (ejection fraction)
   * Radial myocardial velocities
   * Right ventricular function
   * Global diastolic function
   * Left ventricular mass index

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older, men and women, hospitalized and outpatients
* with a history of primary arterial hypertension
* with a daytime ambulatory blood pressure >140 and/or >90 mm Hg
* with left ventricular hypertrophy: LVMI > 125 g/m2 for men, and > 110 g/m2 for women, by Devereux formula, as recommended by the ESH-ESC guidelines (14)
* in sinus rhythm
* consented, by signing the Informed Consent

Exclusion Criteria:

* Severe arterial hypertension (systolic blood pressure > 180 mm Hg and/or diastolic blood pressure > 110 mm Hg)
* Any history of coronary heart disease (stable angina, acute coronary syndromes, myocardial infarction)
* Any history of cerebrovascular disease
* Renal impairment (creatinine > 1.5 mg% for men, > 1.4 mg% for women)
* Left ventricular global systolic dysfunction (EF < 45%)
* More than mild valvar (mitral or aortic) regurgitation
* Hypertrophic cardiomyopathy
* Pericarditis
* Cor pulmonale
* Pregnancy or lactating women
* Any significant co-morbidities
* Contraindication to beta-blocker therapy
* Concomitant treatment with other beta-blockers
* Participation to another investigational study in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-04; Primary Completion 2008-12 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Changes of: longitudinal myocardial velocities at rest (assessed by TDE), systolic functional reserve (calculated as the absolute and relative increase of the myocardial systolic velocities at peak stress from rest), NT-proBNP | 6 months

SECONDARY OUTCOMES:
Global systolic function (ejection fraction) | 6 months
Radial myocardial velocities | 6 months
Right ventricular function | 6 months
Global diastolic function | 6 months
Left ventricular mass index | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dragos VINEREANU, MD, Principal Investigator — University and Emergency Hospital Bucharest, Romania
Locations (1):
- University and Emergency Hospital, Bucharest, Romania

REFERENCES:
- [Derived] Vinereanu D, Madler CF, Gherghinescu C, Ciobanu AO, Fraser AG. Cumulative impact of cardiovascular risk factors on regional left ventricular function and reserve: progressive long-axis dysfunction with compensatory radial changes. Echocardiography. 2011 Sep;28(8):813-20. doi: 10.1111/j.1540-8175.2011.01456.x. Epub 2011 Aug 9. PMID 21827541
- [Derived] Vinereanu D, Gherghinescu C, Ciobanu AO, Magda S, Niculescu N, Dulgheru R, Dragoi R, Lautaru A, Cinteza M, Fraser AG. Reversal of subclinical left ventricular dysfunction by antihypertensive treatment: a prospective trial of nebivolol against metoprolol. J Hypertens. 2011 Apr;29(4):809-17. doi: 10.1097/HJH.0b013e3283442f37. PMID 21297499